CLINICAL TRIAL: NCT01591070
Title: Phase 4 Study of Proactive Treatment of Tacrolimus Ointment for Adult Facial Seborrheic Dermatitis
Brief Title: Proactive Treatment of Tacrolimus Ointment for Adult Facial Seborrheic Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PNUHDM
Record Dates: First submitted 2012-04-25; First posted 2012-05-03 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Seborrheic Dermatitis
Keywords: Facial seborrhoeic dermatitis, tacrolimus
MeSH Terms: conditions — Dermatitis, Seborrheic | interventions — Tacrolimus; Ointments

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- vehicle twice weekly (No Intervention)
- tacrolimus once weekly (Experimental)
  Interventions: Drug: Tacrolimus
- tacrolimus twice weekly (Experimental)
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — 0.1% tacrolimus once-weekly application for 10 weeks
  Other Names: protopic 0.1% ointment
  Arms: tacrolimus once weekly
Drug: Tacrolimus — 0.1% tacrolimus twice weekly application for 10 weeks
  Other Names: protopic 0.1% ointment
  Arms: tacrolimus twice weekly

SUMMARY:
The purpose of this study is to determine whether proactive use of 0.1% tacrolimus ointment once or twice weekly can keep adult facial SD in remission and reduce the incidence of exacerbation.

DETAILED DESCRIPTION:
Seborrhoeic dermatitis (SD) is a common chronic papulosquamous dermatosis, affecting 2% to 10% of the adult population, mainly those between the ages of 20 and 50 years with a male bias. The affected skin appears erythematous and oedematous, covered with yellow-brown scales, and is often accompanied by pruritus. It typically affects areas containing sebaceous glands, particularly the scalp, ears, face, chest, and intertriginous areas. SD has a chronic course, and relapse is common. Therefore, therapy is directed toward reducing the symptoms or aggravating factors of SD, such as loosening and removal of scales and crusts, inhibition of yeast colonization, control of secondary infection, and reduction of erythema and pruritus. Standard topical treatments for SD include corticosteroids and anti-mycotic medications. However, the chronic use of topical corticosteroids particularly on the face could result in undesirable outcomes, such as telangiectasia, atrophy, striae, peri-oral dermatitis, or tachyphylaxis, and early relapse after discontinuation of treatment. SD relapse prevention strategies have not yet been established, so the investigators suspected that intermittent use of tacrolimus ointment can be effective in preventing SD relapse.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age with a diagnosis of facial seborrhoeic dermatitis

Exclusion Criteria:

* taking other systemic or topical treatments for facial seborrhoeic dermatitis within the previous 4 weeks
* a known allergy to the components of tacrolimus ointment
* malignant neoplasm; immunologic abnormality
* active infection
* other definitive cutaneous findings such as erythroderma, acne, and psoriasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2010-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Clinical assessments of erythema, scaling, and pruritus | 12 weeks
  The clinical assessments of erythema, scaling, and pruritus will be evaluated by investigator using 4-point scale: 0 (absent), 1 (mild), 2 (moderate), or 3 (severe).
  Maintenance of stabilised facial Seborroheic dermatitis will be considered those patients who showed significant improvement of clinical assessment in erythema, scaling, and pruritus compared with the baseline values.

CONTACTS AND LOCATIONS:
Overall Officials: Byung-Soo Kim, Ph.D., Study Chair — Pusan National University Hospital
Locations (1):
- Department of dermatology, Pusan National University Hospital, Busan, Busan, South Korea

REFERENCES:
- [Derived] Kim TW, Mun JH, Jwa SW, Song M, Kim HS, Ko HC, Kim MB, Song KH, Lee SK, Seo JK, Lee D, Kim BS. Proactive treatment of adult facial seborrhoeic dermatitis with 0.1% tacrolimus ointment: randomized, double-blind, vehicle-controlled, multi-centre trial. Acta Derm Venereol. 2013 Sep 4;93(5):557-61. doi: 10.2340/00015555-1532. PMID 23388687